CLINICAL TRIAL: NCT04487067
Title: A Phase IIIB, Single Arm, Multicenter Study of Atezolizumab (Tecentriq) in Combination With Bevacizumab to Investigate Safety and Efficacy in Patients With Unresectable Hepatocellular Carcinoma Not Previously Treated With Systemic Therapy-Amethista
Brief Title: A Study of Atezolizumab (Tecentriq) in Combination With Bevacizumab to Investigate Safety and Efficacy in Patients With Unresectable Hepatocellular Carcinoma Not Previously Treated With Systemic Therapy-Amethista
Acronym: AMETHISTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML42243
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab + Bevacizumab (Experimental): Participants will receive atezolizumab 1200 mg intravenous (IV) infusions Q3W (dosed in 3-week cycles) + bevacizumab 15 mg/kg IV Q3W (dosed in 3-week cycles)
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg IV infusion q3w
  Other Names: Tecentriq
Drug: Bevacizumab — Bevacizumab 15 mg/kg IV Q3W
  Other Names: Avastin

SUMMARY:
This is a Phase IIIb, one arm, multicenter, open-label study designed to evaluate the safety and efficacy of atezolizumab + bevacizumab in patients with unresectable HCC who have received no prior systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable HCC with diagnosis confirmed by histology, with a biopsy within 6 months from recruitment;
* Disease that is not amenable to curative surgical and/or locoregional therapies, or progressive disease after surgical and /or locoregional therapies;
* No prior systemic therapy for HCC;
* At least one measurable untreated lesion;
* Patients who received prior local therapy are eligible provided the target lesion(s) have not been previously treated with local therapy or the target lesion(s) within the field of local therapy have subsequently progressed in accordance with RECIST version 1.1;
* ECOG Performance Status of 0 or 1 within 7 days prior to recruitment;
* Child-Pugh class A within 7 days prior to recruitment;
* Patients must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be assessed. In case of varices at high risk of bleeding (corresponding to medium (F2) or large (F3) varices, or F1 varices with cherry red spots or red wale marking) prophylatic treatment per local standard of care must be adopted prior to enrollment. Patients who have undergone an EGD within 6 months of prior to initiation of study treatment do not need to repeat the procedure provided they had no varices at high risk of bleeding;
* Adequate hematologic and end-organ function
* Resolution of any acute, clinically significant treatment-related toxicity from prior therapy to Grade <= 1 prior to study entry, with the exception of alopecia
* Negative HIV test at screening with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥200µL, and have an undetectable viral load;
* In patients with viral HCC, documented virology status of hepatitis, as confirmed by screening HBV and HCV serology test;
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm.

Exclusion Criteria:

* History of leptomeningeal disease or brain metastases;
* Active or history of autoimmune disease or immune deficiency;
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan;
* Known active tuberculosis;
* Significant cardiovascular disease within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina;
* History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death;
* Prior allogeneic stem cell or solid organ transplantation;
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within at least 5 months after the last dose of atezolizumab and 6 months after the last dose of bevacizumab;
* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC;
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high-risk for bleeding;
* A prior bleeding event due to oesophageal and/or gastric varices within 6 months prior to initiation of study treatment;
* Clinically evident ascites;
* Co-infection of HBV and HCV;
* Co-infection with HBV and hepatitis D viral infection;
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases;
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures;
* Clinically significant uncontrolled or symptomatic hypercalcemia;
* Inadequately controlled arterial hypertension;
* Significant vascular disease within 6 months prior to initiation of study treatment;
* History of haemoptysis;
* Evidence of bleeding diathesis or significant coagulopathy;
* History of gastrointestinal (GI) fistula, GI perforation, or intra-abdominal abscess within 6 months prior to initiation of study treatment;
* History of intestinal obstruction and/or clinical signs or symptoms of GI obstruction including sub-occlusive disease related to the underlying disease or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding prior to initiation of study treatment;
* Metastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumor masses of large volume;
* Local therapy to liver within 28 days prior to initiation of study treatment or non-recovery from side effects of any such procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- Italy (21):
  - IRCCS Ospedale Casa Sollievo Della Sofferenza, San Giovanni Rotondo, Apulia
  - Fondazione Pascale, Napoli, Campania
  - Azienda Osp Uni Seconda Università Degli Studi Di Napoli, Napoli, Campania
  - Ospedale del Mare, Napoli, Campania
  - A.O. S. Orsola Malpighi, Bologna, Emilia-Romagna
  - Arcispedale Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - A.O. Universitaria S. Martino Di Genova, Genoa, Liguria
  - Ospedali Riuniti - Bergamo, Bergamo, Lombardy
  - Fondazione IRCCS Ospedale Maggiore Policlinico, Milan, Lombardy
  - Istituto Nazionale Dei Tumori, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Turin, Piedmont
  - A.O.U. Cagliari-P.O. Monserrato, Cagliari, Sardinia
  - A.O.U. Policlinico Paolo Giaccone, Palermo, Sicily
  - Azienda Ospedaliera Di Rilievo Nazionale E Di Alta Specializzazione Garibaldi, Palermo, Sicily
  - A.O.U Careggi, Florence, Tuscany
  - Azlenda Ospendaliero-Universitaria Pisana, Pisa, Tuscany
  - Clinica Oncologica-Ospedali Riuniti Ancona, Torrette, Tuscany
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua, Veneto

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Piscaglia F, Masi G, Martinelli E, Cabibbo G, Di Maio M, Gasbarrini A, Iavarone M, Antonuzzo L, Mazzaferro V, Ballestrero A, Garufi C, Bergamo F, Celsa C, Marino D, Tovoli F, Ponziani FR, Pressiani T, Astolfi C, Gazzoli GC, Ciardiello F, Daniele B, Rimassa L. Atezolizumab plus bevacizumab as first-line treatment of unresectable hepatocellular carcinoma: interim analysis results from the phase IIIb AMETHISTA trial. ESMO Open. 2025 Feb;10(2):104110. doi: 10.1016/j.esmoop.2024.104110. Epub 2025 Jan 27. PMID 39874903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 152 participants with unresectable hepatocellular carcinoma (HCC) and no prior systemic treatment took part in the study at 21 investigative sites in Italy from 25 August 2020 to 13 August 2024.
Pre-assignment Details: Participants received atezolizumab in combination with bevacizumab until unacceptable toxicity or loss of clinical benefit as determined by the investigator. Of the 152 participants enrolled, three participants did not receive any treatment.
Groups:
- Atezolizumab + Bevacizumab: Participants received atezolizumab, 1200 milligrams (mg) as intravenous (IV) infusion, along with bevacizumab, 15 milligrams/kilogram (mg/kg), also as IV infusion, every 3 weeks (Q3W) on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
Period: Overall Study
Arm/Group | Atezolizumab + Bevacizumab
Started | 152
Safety Analysis Population (Safety analysis population included all enrolled participants who had at least one full or partial administration of atezolizumab plus bevacizumab.) | 149
Completed | 21
Not Completed | 131
Not completed — Adverse Event | 3
Not completed — Death Other Than Progressive Disease | 60
Not completed — Death Due To Progressive Disease | 40
Not completed — Lost to Follow-up | 3
Not completed — Progressive Disease | 1
Not completed — Protocol Violation | 3
Not completed — Participant Discontinued From Study as per Protocol | 6
Not completed — Withdrawal by Subject | 15

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who signed the informed consent form (ICF) and were enrolled in the study.
Groups:
- Atezolizumab + Bevacizumab: Participants received atezolizumab, 1200 mg as IV infusion, along with bevacizumab, 15 mg/kg, also as IV infusion, Q3W on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 141
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 145
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3-5 National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE V5) Bleeding/Haemorrhage
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Severity of AEs was graded using NCI CTCAE v5.0. Grade 3=Severe/medically significant but not immediately life-threatening, hospitalization/prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; Grade 4=Life-threatening consequences, urgent intervention indicated; Grade 5=Death related to AE.
Time Frame: Up to approximately 47.6 months
Population: Safety analysis population included all enrolled participants who had at least one full or partial administration of atezolizumab plus bevacizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 149
Participants
  Grade 3 | 17
  Grade 4 | 3
  Grade 5 | 2

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from initiation of study treatment to death from any cause. Kaplan-Meier (K-M) method was used to estimate the OS.
Time Frame: Up to approximately 47.6 months
Population: ITT population included all participants who signed the ICF and were enrolled in the study. Overall number analyzed is the number of participants with data available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 149
months | 20.76 [16.85 to 26.35]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAEs are defined as AEs with onset date on or after the start of the first study treatment component. Number of participants with any TEAEs are reported here.
Time Frame: Up to approximately 47.6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 149
Participants | 144

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from initiation of study treatment to the first occurrence of disease progression (PD) or death from any cause (whichever occurs first), as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1). PD was defined as at least a 20% increase in the sum of diameters (SOD) of target lesions, taking as reference the smallest SOD at prior timepoints (including baseline). In addition to the relative increase of 20%, the SOD must also demonstrate an absolute increase of ≥ 5 millimeters (mm). Participants alive and without any PD were censored at the last assessment date. K-M method was used to estimate the PFS.
Time Frame: Up to approximately 47.6 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 149
months | 8.80 [7.89 to 11.24]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with complete or partial response (CR or PR), as determined by the investigator according to RECIST v1.1. CR was defined as disappearance of all target lesions or any pathological lymph nodes must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR.
Time Frame: Up to approximately 47.6 months
Population: ITT population included all participants who signed the ICF and were enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 152
percentage of participants | 28.29 [0.2173 to 0.3592]

6. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from initiation of study treatment to the first occurrence of PD, as determined by the investigator according to RECIST v1.1. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD at prior timepoints (including baseline). In addition to the relative increase of 20%, the SOD must also demonstrate an absolute increase of ≥ 5 mm. Participants without any PD were censored at the last assessment date. K-M method was used to estimate the TTP.
Time Frame: Up to approximately 47.6 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 149
months | 11.24 [8.48 to 15.77]

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first occurrence of a documented objective response (CR or PR) to PD or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1. CR was defined as disappearance of all target lesions or any pathological lymph nodes must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD at prior timepoints (including baseline). In addition to the relative increase of 20%, the SOD must also demonstrate an absolute increase of ≥ 5 mm. Participants who were alive and without any PD were censored at the last assessment date. K-M method was used to estimate the DOR.
Time Frame: Up to approximately 47.6 months
Population: ITT population included all participants who signed the ICF and were enrolled in the study. Overall number analyzed is the number of participants with an objective response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 43
months | 17.35 [13.54 to 27.24]

8. Secondary Outcome: Post-progression Survival (PPS)
Description: PPS was defined as the time from the first occurrence of PD as determined by the investigator according to RECIST v1.1 to death from any cause. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD at prior timepoints (including baseline). In addition to the relative increase of 20%, the SOD must also demonstrate an absolute increase of ≥ 5 mm. Participants who were alive were censored at the last assessment date. K-M method was used to estimate the PPS.
Time Frame: Up to approximately 47.6 months
Population: ITT population included all participants who signed the ICF and were enrolled in the study. Overall number analyzed is the number of participants with a progressive disease.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 97
months | 11.27 [8.41 to 13.80]

9. Secondary Outcome: Number of Participants Reporting Severe Symptoms in Patient-Reported Outcomes of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Questionnaire
Description: Participants self-reported symptomatic AEs using PRO-CTCAE, a validated item bank used to characterize presence, frequency of occurrence, severity, &/or degree of interference with daily function of 78 patient-reportable symptomatic treatment toxicities. PRO-CTCAE contains questions that are rated either dichotomously (for determination of presence vs. absence) or on a 5-point Likert scale (for determination of frequency of occurrence,severity,& interference with daily function). Treatment toxicities can occur with observable signs (e.g.,vomiting)/ non-observable symptoms (e.g.,nausea). A subset of 14 symptoms most applicable to current treatments were selected for this study. Symptoms were selected based on toxicities associated with the drug's class, mechanism of action, or mode of administration, and toxicities reported with the drug in another indication. Number of participants who reported severe symptoms per the PRO-CTCAE questionnaire on Day 1 of each cycle is reported here.
Time Frame: From Cycle 1 Day 1 to Cycle 63 Day 1 (1 Cycle = 21 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 149
Participants
  Cycle 1 Day 1 | 39
  Cycle 2 Day 1 | 33
  Cycle 3 Day 1 | 23
  Cycle 4 Day 1 | 30
  Cycle 5 Day 1 | 23
  Cycle 6 Day 1 | 22
  Cycle 7 Day 1 | 17
  Cycle 8 Day 1 | 14
  Cycle 9 Day 1 | 19
  Cycle 10 Day 1 | 16
  Cycle 11 Day 1 | 17
  Cycle 12 Day 1 | 16
  Cycle 13 Day 1 | 13
  Cycle 14 Day 1 | 13
  Cycle 15 Day 1 | 9
  Cycle 16 Day 1 | 8
  Cycle 17 Day 1 | 10
  Cycle 18 Day 1 | 10
  Cycle 19 Day 1 | 8
  Cycle 20 Day 1 | 11
  Cycle 21 Day 1 | 5
  Cycle 22 Day 1 | 6
  Cycle 23 Day 1 | 8
  Cycle 24 Day 1 | 10
  Cycle 25 Day 1 | 8
  Cycle 26 Day 1 | 7
  Cycle 27 Day 1 | 8
  Cycle 28 Day 1 | 10
  Cycle 29 Day 1 | 6
  Cycle 30 Day 1 | 7
  Cycle 31 Day 1 | 7
  Cycle 32 Day 1 | 6
  Cycle 33 Day 1 | 6
  Cycle 34 Day 1 | 7
  Cycle 35 Day 1 | 9
  Cycle 36 Day 1 | 8
  Cycle 37 Day 1 | 7
  Cycle 38 Day 1 | 9
  Cycle 39 Day 1 | 8
  Cycle 40 Day 1 | 8
  Cycle 41 Day 1 | 5
  Cycle 42 Day 1 | 6
  Cycle 43 Day 1 | 3
  Cycle 44 Day 1 | 3
  Cycle 45 Day 1 | 3
  Cycle 46 Day 1 | 2
  Cycle 47 Day 1 | 2
  Cycle 48 Day 1 | 3
  Cycle 49 Day 1 | 3
  Cycle 50 Day 1 | 2
  Cycle 51 Day 1 | 3
  Cycle 52 Day 1 | 2
  Cycle 53 Day 1 | 2
  Cycle 54 Day 1 | 1
  Cycle 55 Day 1 | 1
  Cycle 56 Day 1 | 1
  Cycle 57 Day 1 | 0
  Cycle 58 Day 1 | 0
  Cycle 59 Day 1 | 0
  Cycle 60 Day 1 | 0
  Cycle 61 Day 1 | 0
  Cycle 62 Day 1 | 0
  Cycle 63 Day 1 | 0

10. Secondary Outcome: Number of Participants Reporting Very Severe Symptoms in PRO-CTCAE Questionnaire
Description: Participants self-reported symptomatic AEs using PRO-CTCAE, a validated item bank used to characterize presence, frequency of occurrence, severity, &/or degree of interference with daily function of 78 patient-reportable symptomatic treatment toxicities. PRO-CTCAE contains questions that are rated either dichotomously (for determination of presence vs. absence) or on a 5-point Likert scale (for determination of frequency of occurrence,severity,& interference with daily function). Treatment toxicities can occur with observable signs (e.g.,vomiting)/ non-observable symptoms (e.g.,nausea). A subset of 14 symptoms most applicable to current treatments were selected for this study. Symptoms were selected based on toxicities associated with the drug's class, mechanism of action, or mode of administration, &toxicities reported with the drug in another indication. Number of participants who reported very severe symptoms per the PRO-CTCAE questionnaire on Day 1 of each cycle is reported here.
Time Frame: From Cycle 1 Day 1 to Cycle 63 Day 1 (1 Cycle = 21 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 149
Participants
  Cycle 1 Day 1 | 15
  Cycle 2 Day 1 | 18
  Cycle 3 Day 1 | 12
  Cycle 4 Day 1 | 12
  Cycle 5 Day 1 | 10
  Cycle 6 Day 1 | 11
  Cycle 7 Day 1 | 7
  Cycle 8 Day 1 | 11
  Cycle 9 Day 1 | 7
  Cycle 10 Day 1 | 7
  Cycle 11 Day 1 | 6
  Cycle 12 Day 1 | 5
  Cycle 13 Day 1 | 7
  Cycle 14 Day 1 | 7
  Cycle 15 Day 1 | 7
  Cycle 16 Day 1 | 8
  Cycle 17 Day 1 | 4
  Cycle 18 Day 1 | 5
  Cycle 19 Day 1 | 4
  Cycle 20 Day 1 | 4
  Cycle 21 Day 1 | 1
  Cycle 22 Day 1 | 4
  Cycle 23 Day 1 | 2
  Cycle 24 Day 1 | 3
  Cycle 25 Day 1 | 4
  Cycle 26 Day 1 | 4
  Cycle 27 Day 1 | 3
  Cycle 28 Day 1 | 3
  Cycle 29 Day 1 | 3
  Cycle 30 Day 1 | 2
  Cycle 31 Day 1 | 4
  Cycle 32 Day 1 | 3
  Cycle 33 Day 1 | 3
  Cycle 34 Day 1 | 5
  Cycle 35 Day 1 | 5
  Cycle 36 Day 1 | 3
  Cycle 37 Day 1 | 6
  Cycle 38 Day 1 | 4
  Cycle 39 Day 1 | 4
  Cycle 40 Day 1 | 4
  Cycle 41 Day 1 | 4
  Cycle 42 Day 1 | 5
  Cycle 43 Day 1 | 4
  Cycle 44 Day 1 | 4
  Cycle 45 Day 1 | 2
  Cycle 46 Day 1 | 2
  Cycle 47 Day 1 | 1
  Cycle 48 Day 1 | 1
  Cycle 49 Day 1 | 0
  Cycle 50 Day 1 | 1
  Cycle 51 Day 1 | 0
  Cycle 52 Day 1 | 1
  Cycle 53 Day 1 | 1
  Cycle 54 Day 1 | 0
  Cycle 55 Day 1 | 1
  Cycle 56 Day 1 | 0
  Cycle 57 Day 1 | 1
  Cycle 58 Day 1 | 0
  Cycle 59 Day 1 | 0
  Cycle 60 Day 1 | 0
  Cycle 61 Day 1 | 0
  Cycle 62 Day 1 | 0
  Cycle 63 Day 1 | 0

11. Other Pre Specified Outcome: Number of Participants Starting Second or Further Lines of Treatment
Time Frame: Up to approximately 47.6 months
Population: Per protocol, this is an exploratory outcome measure; therefore, the results have not been reported.
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Other AEs: From initiation of study drug until 30 days after the final dose or initiation of new systemic anti-cancer therapy, whichever occurs first (up to approximately 47.6 months) SAEs, and All-cause mortality: From initiation of study drug until 90 days after the final dose or initiation of new systemic anti-cancer therapy, whichever occurs first (up to approximately 47.6 months)
Description: Safety analysis population included all enrolled participants who had at least one full or partial administration of atezolizumab plus bevacizumab.
Arm/Group | Atezolizumab + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 102/149
Serious Adverse Events (participants affected / at risk) | 62/149
Other Adverse Events (participants affected / at risk) | 142/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab + Bevacizumab (N=149)
Anaemia (Blood and lymphatic system disorders) | 3 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (5)
Myocardial infarction (Cardiac disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 3 (3)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 4 (4)
Pancreatic haemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3)
Chest pain (General disorders) | 1 (2)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Biliary tract infection (Infections and infestations) | 2 (2)
Brain abscess (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Peri-implantitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 5 (5)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Electrocardiogram abnormal (Investigations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Hepatic encephalopathy (Nervous system disorders) | 2 (2)
Hypoglycaemic coma (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (3)
Confusional state (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Leg amputation (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 2 (2)
Pelvic venous thrombosis (Vascular disorders) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab + Bevacizumab (N=149)
Asthenia (General disorders) | 64 (97)
Pyrexia (General disorders) | 32 (38)
Fatigue (General disorders) | 26 (30)
Oedema peripheral (General disorders) | 12 (14)
Mucosal inflammation (General disorders) | 10 (12)
Hypertension (Vascular disorders) | 51 (99)
Diarrhoea (Gastrointestinal disorders) | 42 (64)
Abdominal pain (Gastrointestinal disorders) | 25 (32)
Nausea (Gastrointestinal disorders) | 22 (28)
Ascites (Gastrointestinal disorders) | 16 (18)
Abdominal pain upper (Gastrointestinal disorders) | 14 (16)
Constipation (Gastrointestinal disorders) | 14 (16)
Vomiting (Gastrointestinal disorders) | 14 (15)
Stomatitis (Gastrointestinal disorders) | 10 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 36 (46)
Decreased Appetite (Metabolism and nutrition disorders) | 33 (42)
Proteinuria (Renal and urinary disorders) | 28 (48)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (43)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (29)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (23)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Headache (Nervous system disorders) | 18 (21)
Hypothyroidism (Endocrine disorders) | 17 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (35)
Anaemia (Blood and lymphatic system disorders) | 15 (17)
Blood bilirubin increased (Investigations) | 13 (21)
Platelet count decreased (Investigations) | 11 (19)
Aspartate aminotransferase increased (Investigations) | 11 (14)
Alanine aminotransferase increased (Investigations) | 8 (10)
COVID-19 (Infections and infestations) | 13 (14)
Hypertransaminasaemia (Hepatobiliary disorders) | 9 (13)
Hyperbilirubinaemia (Hepatobiliary disorders) | 8 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT04487067/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT04487067/SAP_001.pdf